CLINICAL TRIAL: NCT03266250
Title: Transthoracic Echocardiography of Inferior Vena Cava Before Spinal Anesthesia Can Predict Hypotension in Elderly Orthopaedic Patients
Brief Title: Transthoracic Echocardiography of Inferior Vena Cava Before Spinal Anesthesia Can Predict Hypotension
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Theodosis Saranteas, MD, Assistant Professor, National and Kapodistrian University of Athens
Other Study IDs: ED399,09-24-2015
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2017-08

CONDITIONS: Spinal Anesthetic Toxicity; Inferior Vena Cava Abnormality; Intraoperative Complications
Keywords: inferior vena caca ultrasound
MeSH Terms: conditions — Intraoperative Complications | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spinal anesthesia Hypotensive patients: Transthoracic echocardiography of IVC before spinal anaesthesia
  Interventions: Procedure: spinal anesthesia
- spinal anesthesia Normotensive patients: Transthoracic echocardiography of IVC before spinal anaesthesia
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Transthoracic echocardiography of inferior vena cava before spinal anesthesia

SUMMARY:
Study Protocol: Outcome Measurements Primary Outcome The main outcome will be the preoperative performance of the dIVCmax/IVCCI ratio to foresee the incidence of hypotension after spinal anesthesia in a greater extent to that of the established IVCCI measurements.

Secondary Outcomes To identify other echocardiographic or clinical measurements that can predict an intraoperative spinal-induced haemodynamic instability.

Sample Size Calculation A pilot study of 20 patients revealed a detected area under the ROC curve (AUC) of 0,91 for dIVCmax/IVCCI and for dIVCmax 0,82 with rank correlation between the two assays being 0.87 in both positive and negative cases. Based on this result, a sample of 56 patients will achieve 80% power to detect significant difference (at a level 0.05) between dIVCmax/IVCCI and dIVCmax.

Potential Benefits of the Study The results of this study will allow us to determine which clinical or US-measurement can yield better performance so as a preoperative prediction of spinal-induced hypotension can be achieved; that way these measurements can permit and guide a targeted preoperative fluid challenges prior to the implementation of spinal anesthesia Potential Side Effects of the Study Participation in this protocol will not put patients at higher risk for complications since we do not perform any intervention (either pharmacological or surgical) There will be no occupational risks to researchers or assistants. Proposed Timetable According to the exclusion criteria and taking into account the number of cases performed in our department per monthly basis, it should take us approximately 6 months to recruit 60 patients.

DETAILED DESCRIPTION:
AIM OF THE STUDY

We hypothesized, therefore, that the preoperative dIVCmax/IVCCI ratio (maximum diameter of inferior vena cava-IVC- at the expiration = dIVCmax and the collapsibility index of the IVC =IVCCI) could greater foresee the incidence of hypotension after spinal anesthesia than the established IVCCI measurements. In light of this hypothesis, we prospectively examined both the dIVCmax/IVCCI ratio and IVCCI before spinal anesthesia in a population who fulfilled predetermined inclusion criteria and we set out to evaluate the diagnostic performance of this indices in predicting spinal-induced hypotension.

METHODOLOGY In the present observational prospective study, consecutive sampling is used to recruit ageing patients (>70 years) who sustained orthopaedic operation under spinal anesthesia.

According to our department policy, the documentation of a cardiac disease in our patients takes place during the routine preoperative anesthetic evaluation always with the cooperation of consultant cardiologists. Patients' medical history, physical examination, ECG, and X-ray assessment are standard practice supplemented by specific exams or tests Echocardiogrphic protocol and measurements A TTE is performed in all patients before spinal anaesthesia (Vivid T8, GE Healthcare, Waukesha, Wisconsin, USA) equipped with a 2-5 MHz phased array transducer. All echocardiograms is carried out by the same anesthesiologist/intensivist (TS), who has 12 years of experience in perioperative echocardiography. All data are saved and stored digitally for off-line analysis.

A standard intraoperative TTE protocol is being used in all patients. and included the following views: subxiphoid4-chamber (SUBX), apical 4-chamber (4CH), apical 2-chamber (2CH), apical 3-chamber (3CH), parasternal long (LAX) and short axis (SAX) windows.

All data are saved and stored digitally for off-line postoperative analysis. The Ejection Fraction (EF) is determined using the Simpson's method. Patients with EF lower than 50% do not continue for the study. The global longitudinal peak systolic strain (GLPSS) is used to assess LV mechanics in the longitudinal axis of LV motion. The TAPSE index is employed for the assessment of the right ventricular function. LV filling pressures in diastole is estimated by the E/Em ratio (E=peak velocity flow in early diastole, Em=the average of peak velocities in early diastole of lateral and septal mitral annulus). In addition, LV dimensions and wall thickness are measured either in short or long parasternal axis view. Stroke volume of the LV is assessed by VTILVOT (pulsed-wave Doppler of velocity time integral in the LV outflow tract).

IVC measurements included its maximum diameter at the end of expiration (dIVCmax), IVCCI during spontaneous in quite breathing, [(IVC maximal diameter - IVC minimal diameter)/IVC maximal diameter] and the ratio (R) of dIVCmax/IVCCI; the IVC diameters were measured in the long axis of the IVC and just proximal to the entry of the hepatic veins.

Anesthetic protocol and measurements. Spinal anaesthesia is introduced with a single intrathecal injection of 0.75% plain ropivacaine using a 22 or 25-gauge needle with the patient in the lateral or sitting position. The dose range is 12mg to 18mg, depending on age and height. Perioperative hemodynamic monitoring is carried out with an indwelling radial artery catheter. Patients with intraoperative mean blood pressure (MBP) ≤65 mmHg, or <25% of its baseline preoperative value were considered hypotensive. Arterial hypotension related to bone cement application, tourniquet deflation, overt intraoperative/postoperative bleeding (blood loss>150cc) or patients receiving blood transfusion for any reason were not considered.

Statistical analysis Sample size: A pilot study of 20 patients revealed a detected area under the ROC curve (AUC) of 0,91 for dIVCmax/IVCCI and for dIVCmax 0,82 with rank correlation between the two assays being 0.87 in both positive and negative cases. Based on this result, a sample of 56 patients achieved 80% power to detect significant difference (at a level 0.05) between dIVCmax/IVCCI and dIVCmax.

Data analysis: Quantitative variables and proportions will be compared with the student t-test and chi-square test respectively. Normality was tested by using the Kolmogorov-Smirnov test. Receiver operating characteristic (ROC) curve analysis will be performed to evaluate the diagnostic performance of clinical/Doppler parameters in identifying patients who experienced spinal-induced hypotension. The area under the curve (AUC) and the respective 95% confidence interval (95% CI) are estimated according to Hanley and McNeil. 1 The AUC curves are compared using the method described by DeLong et al. 2. The results are expressed as percentage (%) or mean ± SD; a p value of <0.05 is considered statistically significant. Statistical analysis will be done with statistical analysis software (SPSS, 17.0, Chicago, IL; MedCalc Software, Mariakerke, Belgium).

1. Hanley JA, McNeil BJ. The meaning and use of the area under a receiver operating characteristic (ROC) curve. Radiology 1982 ;143:29-36
2. DeLong ER, DeLong DM, Clarke- Pearson DL. Comparing the areas under two or more correlate receiver operating characteristic curves: a nonparametric approach. Biometrics 1988; 44:837-845

ELIGIBILITY:
Inclusion Criteria: patients with AHA/ACC stage I, II or III with their cardiac disease status in compensated status -

Exclusion Criteria: patients with AHA/ACC stage IV

-

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly orthopaedic patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Preoperative performance of the dIVCmax/IVCCI ratio | 6 months
  The main outcome will be the preoperative performance of the dIVCmax/IVCCI ratio to foresee the incidence of hypotension after spinal anesthesia in a greater extent to that of the established IVCCI measurements

SECONDARY OUTCOMES:
Echocardiographic or clinical measurements | 6 months
  To identify other echocardiographic or clinical measurements that can predict an intraoperative spinal-induced haemodynamic instability

CONTACTS AND LOCATIONS:
Overall Officials: Theodosis Saranteas, MD, Principal Investigator — National and Kapodistrian University of Athens, School of Medicine
Locations (1):
- ATTIKON University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang J, Critchley LA. Inferior Vena Cava Ultrasonography before General Anesthesia Can Predict Hypotension after Induction. Anesthesiology. 2016 Mar;124(3):580-9. doi: 10.1097/ALN.0000000000001002. PMID 26771910